CLINICAL TRIAL: NCT06105112
Title: Minimally Invasive Periodontal Regeneration With a Combination Approach Using Either Hyaluronic Acid or Enamel Matrix Derivatives: a 24-month Multicenter Randomized Controlled Clinical Trial
Brief Title: Periodontal Regeneration With Hyaluronic Acid or Enamel Matrix Derivatives
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Aimetti, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HATurin
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic acid (Experimental): Minimally invasive surgical technique with a combined approach using hyaluronic acid gel and a bone xenograft.
  Interventions: Device: Hyaluronic acid
- Enamel matrix derivatives (Active Comparator): Minimally invasive surgical technique with a combined approach using enamel matrix derivatives gel and a bone xenograft.
  Interventions: Device: Enamel matrix derivatives

INTERVENTIONS:
Device: Hyaluronic acid — Minimally invasive flap elevation and debridement of the intrabony defect with micro-curettes. Root surface debridement with ultrasonic debridement with periotip and mini-curettes. Application of cross-linked hyaluronic acid gel composed of a mixture of cross-linked (1.6%) and natural (0.2%) hyaluronic acid (hyaDent BG, Regedent, Germany) through a syringe over a bone xenograft (Smartgraft, Regedent, Germany). The mixture will be then compacted within the intrabony component of the defect.
  Arms: Hyaluronic acid
Device: Enamel matrix derivatives — Minimally invasive flap elevation and debridement of the intrabony defect with micro-curettes. Root surface debridement with ultrasonic debridement with periotip and mini-curettes. Enamel matrix derivatives gel (Emdogain, Straumann, Switzerland) will be applied on the dry root surfaces and left in place for at least 1 minute avoiding blood contamination. Subsequently, a bone xenograft (Smartgraft, Regedent, Germany) will be compacted within the intrabony component of the defect.
  Arms: Enamel matrix derivatives

SUMMARY:
To date, the quest for ideal biological inductors for periodontal regeneration is still ongoing, especially when facing non-containing defect anatomies. The primary aim of this study is to evaluate the clinical and radiographic performance of a bone graft combined with either enamel matrix derivatives or hyaluronic acid for periodontal regeneration of non-containing intrabony defects in terms of clinical attachment gain (primary outcome) and other secondary outcomes (probing pocket depth reduction, radiographic bone fill). Moreover, this study aims to compare early wound healing and patient-reported outcome measures.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of stage III-IV periodontitis.
* Completed steps I-II periodontal therapy.
* FMPS <15% at 3-month re-evaluation.
* FMBS <15% at 3-month re-evaluation.
* At least one site with intrabony defects and residual PPD ≥ 6 mm at re-evaluation, with a radiographic intrabony component ≥ 3 mm, and limited to no extension of the defect on the lingual or palatal side as assessed by preoperative bone sounding.
* Intrasurgically, the defect has to present a non-supporting anatomy (1-2 residual walls in its most coronal portion) and it needs to be accessible by flap elevation only on one side (either buccal or oral).
* Signed informed consent.

Exclusion criteria:

* Compromised general health which contraindicates the study procedures (ASA III-VI patients).
* Systemic diseases/medications which could influence the outcome of the therapy (e.g. uncontrolled diabetes mellitus, non-plaque-induced gingival diseases, antiepileptic drugs (phenytoin and sodium valproate), certain calcium channel-blocking drugs (e.g., nifedipine, verapamil, diltiazem, amlodipine, felodipine), immunoregulating drugs (e.g., ciclosporine), and high-dose oral contraceptives).
* Current smokers (self-reported, ≥ 10 cigarettes a day), users of chewing tobacco, and drug/alcohol abusers.
* Pregnant or nursing women.
* Presence of furcation involvement ≥ II degree (Hamp 1975) at the affected teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level change | 24 months
  Clinical attachment level will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

SECONDARY OUTCOMES:
Probing pocket depth change | 24 months
  Probing depth will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)
Radiographic bone level change | 24 months
  Periapical standardized radiographs will be taken by a clinician masked to the clinical measurements using the paralleling technique and individually customized bite-blocks (RINN XCP Film Holding Instruments, Dentsply, York, USA)
Patient reported outcome measures | 14 weeks
  Pain will be self-recorded by the patient using a visual analog scale (from 0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy